CLINICAL TRIAL: NCT07221825
Title: Low-Count Quantitative SPECT for Men Treated With Radium-223
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202506234; R01EB031962 (NIH)
Record Dates: First submitted 2025-10-25; First posted 2025-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Cancer of the Prostate
Keywords: Prostate cancer; Bone metastasis; SPECT; Radiopharmaceutical therapies; Theranostics; Alpha-particle; Xofigo
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LC-QSPECT (Experimental): Consenting and eligible men receiving standard of care (Xofigo) will receive a noninvasive LC-QSPECT scan (~45 minutes) and a low-dose contrast-enhanced CT after Cycles 1 and 3 of Xofigo. SOC CT and bone scans will also be performed at baseline and after Cycles 3 and 6. Specimen collection will be as follows: bone biopsy (Cycle 1 Day 2) (optional), stool (first bowel movement post-each SPECT scan), and blood for PSA and bone turnover biomarkers (with each cycle of treatment). Additionally, pain will be assessed, and quality of life will be monitored prior to treatment and after each treatment cycle.
  Interventions: Device: Low-count quantitative single-photon emission computed tomography imaging
- Physicians (No Intervention): Additionally, medical oncologists and radiation oncologists who are seeing patients who are enrolled in this study will be considered participants in this study (as they will be completing the Physician Questionnaire).

INTERVENTIONS:
Device: Low-count quantitative single-photon emission computed tomography imaging — LC-QSPECT scans will be performed between 6 and 36 hours after administration of Xofigo during Cycles 1 and 3.
  Other Names: LC-QSPECT
  Arms: LC-QSPECT

SUMMARY:
Internal radiotherapies (radiolabeled molecules that are systemically administered and localize to sites of disease) provide cancer-ablating doses to diseased cells while sparing adjacent normal tissues. [223Ra]RaCl2 (Xofigo) is the first FDA-approved alpha-particle emitting radiopharmaceutical therapy (αRPT), providing a survival benefit for men with bone metastatic castration-resistant prostate cancer. Systemically administered radiotherapies distribute throughout the patient, accumulating to unknown levels at sites of disease and in radiosensitive vital organs. The whole-body distribution means that absorbed doses in the patient extend far beyond a pre-defined treatment field. There is a lack of information about αRPT distribution and localization, and this confounds treatment monitoring, complicates dose and schedule personalization, and impedes drug development.

Single-photon emission computed tomography (SPECT) imaging offers a mechanism to quantify uptake; however, αRPT administered activities are significantly lower than those used with diagnostic procedures, which presents a challenge for quantitation with conventional methods. Preliminary research shows that low-count quantitative SPECT (LC-QSPECT) imaging demonstrates reliable quantitation of regional uptake for αRPTs. The purpose of this study is to demonstrate the feasibility, tolerability and performance of LC-QSPECT imaging.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Histologically or cytologically confirmed castration-resistant prostate cancer with symptomatic bone metastases.
* Minimum detectable skeletal lesion count of 3.
* Eligible to receive Xofigo.
* At least 18 years of age.
* ECOG performance status ≤ 3.
* Ability to understand and willingness to sign an IRB-approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria - Patients:

* Predominant visceral metastatic disease.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Concurrent alternative radiopharmaceuticals
* Inability to maintain stationary supine pose for 45-60 minutes

Eligibility Criteria - Physicians:

* Medical Oncologist or Radiation Oncologist at Siteman Cancer Center.
* Treating patients with prostate cancer.
* Willing to complete Physician Questionnaire during participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Spearman's correlation coefficient between the LC-QSPECT estimated uptake in the lesions and intestine with ex vivo activity sampling | Through collection of ex vivo sample (estimated to be 3 months)
  The investigators will assess if the correlation (in absolute magnitude) ≥ 0.60 between the tissue and SPECT data against a low correlation of < 0.2 based on 1-sided normal test at a 5% level.

SECONDARY OUTCOMES:
LC-QSPECT related adverse events | From start of LC-QSPECT imaging through 12 hours following LC-QSPECT imaging
Percentage of enrolled patients who withdraw from the study due to adverse events at least possibly related to LC-QSPECT (as chosen by patients or treating physician team) | From start of LC-QSPECT imaging through 12 hours following LC-QSPECT imaging
Feasibility of conducting LC-QSPECT will be determined by percentage of SPECT scans that can be processed using the investigators' computational method | Through completion of LC-QSPECT imaging (estimated to be 3 months)
  Feasibility is defined as at least 80% of scans able to be processed.
Correlation between the LC-QSPECT measurements and PSA (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
Correlation between the LC-QSPECT measurements and PSA doubling time (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
Correlation between the LC-QSPECT measurements and bone-turnover markers (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
Correlation between the LC-QSPECT measurements and Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  * Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
  * The FACT-P scale is a tool used for assessing the health-related quality of life (QoL) in men with prostate cancer. It consists of 27 core items which assess patient function in four domains (Physical, Social/Family, Emotional, and Functional well-being), and it is further supplemented by 12 site specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce a global QoL score, with a range of scores of 0 to 156. Higher scores represent better QoL.
Correlation between the LC-QSPECT measurements and EuroQol-5 (EQ-5D-5L) questionnaire (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  * Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
  * EQ-5D-5L is a descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension. Scale Minimum: 0. Scale Maximum: 100. Higher score indicates better outcome.
Correlation between the LC-QSPECT measurements and Brief Pain Inventory (BPI) questionnaire (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  * Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
  * BPI score ranges from 0 to 10 with a higher score denoting a higher pain severity.
Correlation between the LC-QSPECT measurements and bone turnover (Spearman Correlation Coefficient) | Through completion of Xofigo treatment (estimated to be 6 months)
  Spearman correlation coefficient measures the strength and direction of the linear correlation (dependence) between 2 variables after converting the raw data to ranks, giving a value between +1 and -1 inclusive, where 1 indicates perfect positive correlation, 0 indicates no correlation, and -1 indicates perfect negative correlation.
Percentage of times that the use of the LC-QSPECT procedure resulted in any changes in treatment plans of the patients | Through completion of Xofigo treatment (estimated to be 6 months)
Performance of the LC-QSPECT procedure using a no-gold-standard evaluation technique. | Through completion of LC-QSPECT imaging (estimated to be 3 months)
  * The investigators will use the no-gold-standard technique to assess whether the LC-QSPECT technique yields precise performance on the task of isotope uptake quantification, where slope and noise will be estimated and the noise-to-slope ratio (NSR) will be calculated.
  * The no-gold-standard technique can be found here: Jha AK, Caffo B, Frey EC. A no-gold-standard technique for objective assessment of quantitative nuclear-medicine imaging methods. Phys Med Biol. 2016 Apr 7;61(7):2780-800. doi: 10.1088/0031-9155/61/7/2780. Epub 2016 Mar 16. PMID: 26982626; PMCID: PMC4921224 and here: Yan Liu, Ziping Liu, Zekun Li, Daniel Thorek, Barry Siegel, Abhinav Jha, "No-gold-standard evaluation of quantitative SPECT methods for alpha-particle radiopharmaceutical therapy", Journal of Nuclear Medicine Jun 2023, 64 (supplement 1) P1331

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav K Jha, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified SPECT imaging data, quantitative imaging metrics, and limited clinical variables (e.g., demographics, treatment cycle, administered activity, relevant lab values, clinical outcome measures) may be shared with qualified researchers at academic, nonprofit, or industry institutions for secondary analyses of image data, dosimetry, quantitative modeling, or clinical outcomes related to Radium-223 therapy.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months after publication of primary results; available for at least 5 years.
Access Criteria: Data will be shared through a controlled-access repository. Access will require a brief proposal and a signed data use agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu